CLINICAL TRIAL: NCT05713630
Title: TRACE STUDY: A Randomized Controlled Trial Using Tranexamic Acid in the Treatment of Subdural Hematoma
Brief Title: The Use of Tranexamic Acid in the Treatment of Symptomatic Subdural Hematoma
Acronym: TRACE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 471164
Record Dates: First submitted 2023-01-26; First posted 2023-02-06 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Subdural Hematoma
Keywords: symptomatic subdural hematoma; tranexamic acid; TXA; clinical trial; neurosurgery
MeSH Terms: conditions — Hematoma, Subdural | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Vanguard trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Research Assistant Research Coordinator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard care + TXA (Active Comparator): Patients will be given a single oral or IV loading dose of TXA within three hours of being randomized or whenever possible prior to surgery. Patients who are able to swallow will be given an oral loading dose of 1g TXA. Patients who are unable to swallow will be given an IV loading dose of 1g TXA which will be added to a 100mL infusion bag of NaCl 0.9% and infused by slow intravenous injection over 20 minutes as per the recommended rate of administration in the Product Monograph for Sandoz-Tranexamic Acid Injection BP. After 12 hours of the loading dose, patients will be given 500mg TXA by mouth (or 500mg TXA in NaCl 0.9% 100mL by IV for those unable to swallow) three times daily, totalling 1500mg/day, for 45 days.
  Interventions: Drug: Tranexamic acid (TXA)
- Standard care + placebo (Placebo Comparator): Patients will be given a single oral or IV loading dose of placebo within three hours of being randomized or whenever possible prior to surgery. Patients who are able to swallow will be given an oral loading dose of 1g placebo (gelatin capsule composed of microcrystalline cellulose 105 powder NF). Patients who are unable to swallow will be given an IV loading dose of 1g placebo (sodium chloride also known as NaCl 0.9%) which will be added to a 100mL infusion bag of NaCl 0.9% and infused by slow intravenous injection over 20 minutes. After 12 hours of the loading dose, patients will be given 500mg placebo by mouth (or IV for those unable to swallow) three times a day, totalling 1500mg/day, for 45 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic acid (TXA) — Marcan-Tranexamic Acid 500 mg oral tablet over-encapsulated to match the placebo. Sandoz-Tranexamic Acid 100 mg/mL solution for injection via intravenous (IV) added to a 100mL infusion bag of NaCl 0.9% and infused by slow intravenous injection over 20 minutes.
  Other Names: Cyklokapron
  Arms: Standard care + TXA
Drug: Placebo — Placebo 500 mg consisting of an identical capsule to over-encapsulated tranexamic acid oral tablet entirely filled with microcrystalline cellulose, and sealed. Placebo 100 mg/mL solution for injection via intravenous (IV) consisting of 0.9% sodium chloride (saline).
  Arms: Standard care + placebo

SUMMARY:
Subdural hematoma (SDH) is a common condition experienced after head injury. Blood collects on the surface of the brain, causing headaches which can progress to confusion, weakness, or even coma. While patients with SDH often receive surgery, not all patients require surgery right away to ease pressure on the brain. After surgery, there can be up to 30 percent chance of more bleeding and the need for more surgeries. Given this, a drug capable of lowering the chance of more bleeding and speeding the recovery of the patient is highly desirable. In this study, we will test a commonly used, cheap drug called Tranexamic Acid (TXA). While the body stops unwanted and sometimes dangerous bleeding naturally by forming blood clots, TXA stops these blood clots from breaking down, which helps to keep bleeding spots plugged. Our previous study showed that TXA helped speed up patients' recovery; but a larger number of patients is necessary to evaluate how well TXA works to reduce bleeding and improve patient-reported outcomes. In this study, regardless of the need for surgery, half of the patients will be randomly assigned to take TXA, while the other half will take a placebo, which is a look-alike substance that contains no active drug. We will measure multiple outcomes over time to determine if TXA is working and lowers healthcare and personal costs, while also taking blood and surgical samples, to better understand how this drug works in SDH patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 45 and older weighing between 45-150 kg diagnosed with symptomatic SDH will be included. SDH is defined as unilateral or bilateral crescentic collection of blood (hyper, iso, or hypodense, or mixed density) of greater than or equals to 8 mm in thickness along the cerebral convexity on CT of the head. Symptomatic SDH patients eligible for inclusion are those with SDH with one or more of the following symptoms attributable to the SDH: headache, gait disturbance, confusion or cognitive decline, limb weakness or numbness/paresthesia, speech or visual disturbance, drowsiness or impaired consciousness, seizures, impaired cognition, or memory loss at the time of assessment.

Exclusion Criteria:

- Patients will be excluded for any of the following conditions:

1. Asymptomatic for longer than 72 hours
2. SDH less than 8 mm in maximal thickness
3. Have an acutely deteriorating neurological status (e.g., brain herniation with pupillary dilation, aneurysm rupture, etc.) that is likely to be fatal within 6 hours or less due to a predominantly acute SDH
4. Presence of brain contusion larger than 5 cubic centimeters or subarachnoid hemorrhage (SAH) thicker than 10 mm with Glasgow Coma Scale (GCS)< 13
5. Patients with primarily interhemispheric or tentorial SDH
6. Hypersensitivity to TXA or any of the placebo ingredients
7. Pregnancy
8. Irregular menstrual bleeding with unidentified cause
9. Known acquired colour vision disturbances
10. Hematuria caused by renal parenchymal disease
11. Acute and chronic renal insufficiency indicated by estimated Glomerular Filtration Rate (eGFR) ≤ 30 mL/min
12. Concomitant intake of birth control pill and/or hormonal replacement therapy, and anti-inhibitor coagulant concentrates (factor VIII inhibitor bypass activity (FEIBA), factor VII, activated factor IX)
13. Consumption coagulopathy/disseminated intravascular coagulation (DIC) in the last 7 days
14. Not competent to take study medication properly and regularly or not having access to caregiver that is able to comply with study medication administration
15. Mechanical heart valve
16. Liver cirrhosis
17. Recent venous and/or arterial thromboembolism within 6 months of study enrolment
18. SDH caused by intracranial hypotension
19. Known thrombophilia (e.g., antiphospholipid syndrome)
20. Any active malignancy: metastatic cancer systemically or to the brain or a primary malignant brain tumour treated within the last 6 months
21. Previous enrolment in this trial for a prior episode
22. Time interval >3 days from the time of clinical assessment to eligibility assessment
23. Patients weighing <45 kg or >150 kg

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2027-03-30 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
European Quality of Life 5 Dimensions 5 Level Version (EQ-5D-5L) | Every 2 weeks after randomization up to 45±10 days.
  A self-rated questionnaire that assesses a patient's health state in five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) Scale v1.2 - Global Health. English and French versions | Baseline and every 2 weeks after randomization up to 45±10 days, and then at 60-90 days, and 180±10 days after randomization.
  A 10-item measure that assesses an individual's general physical, mental, and social health as it is intended to globally reflect individuals' assessment of their physical and mental health in the last 7 days.
PROMIS Item Bank v2.0 - Cognitive Function. English version | Baseline and every 2 weeks after randomization up to 45±10 days, and then at 60-90 days, and 180±10 days after randomization.
  A measure that assesses cognitive function that will be administered as a computer adaptive test.
PROMIS Item Bank v2.0 - Physical Function. English version | Baseline and every 2 weeks after randomization up to 45±10 days, and then at 60-90 days, and 180±10 days after randomization.
  A measure that assesses self-reported capability rather than actual performance of physical activities that will be administered as a computer adaptive test.
PROMIS Item Bank v2.0 - Ability to Participate in Social Roles and Activities. English version | Baseline and every 2 weeks after randomization up to 45±10 days, and then at 60-90 days, and 180±10 days after randomization.
  A measure that assesses the perceived ability to perform one's usual social roles and activities that will be administered as a computer adaptive test. The item bank does not use a time frame (e.g. over the past 7 days) when assessing ability to participate in social roles and activities.
Subdural hematoma volume change | Baseline, 45±10 days after randomization, and 60-90 days if deemed necessary for the patient's routine care.
  Change in hematoma volume in millilitres on CT scan.
Number of subdural hematoma-related surgical interventions | First admission, subsequent admissions up to 180 days after randomization
Recurrence rate of SDH | 45±10 days, 60-90 days, and 180±10 days after randomization
Mortality | During the course of study up to 180±10 days after randomization
Modified Rankin Scale | Baseline, 45±10 days, 60-90 days, and 180±10 days after randomization
  A 6-point disability scale used to measure the degree of disability in patients who have had a stroke.
Disability Rating Scale | Baseline, 45±10 days, 60-90 days, and 180±10 days after randomization
  Eight questions regarding body function, activity, participation, communication, and movements each rated on a 3-5-point scale that is summed to give a total score.
Montreal Cognitive Assessment | Baseline, 45±10 days, and 60-90 days after randomization
  This assessment evaluates the patient's cognition based on eight areas: visuospatial/executive function, naming, memory, attention, language, abstraction, delayed recall, and orientation.
Medical Consumption Questionnaire | Baseline, 45±10 days, and 180±10 days after randomization
  Health-related cost questionnaire on the use of healthcare in the past month.
EQ-5D-5L | Baseline, 60-90 days, and 180±10 days after randomization
  A self-rated questionnaire that assesses a patient's health state in five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Adverse events | Discharge, 45±10 days, 60-90 days, and 180±10 days after randomization
  Adverse events of grade 3 or higher as defined by Good Clinical Practice Guidelines.
Length of stay in hospital due to subdural hematoma | During the course of the study up to 180±10 days after randomization
Disposition after discharged from hospital | During the course of the study up to 180±10 days after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Cusimano, MD, PhD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fu TS, Jing R, McFaull SR, Cusimano MD. Recent trends in hospitalization and in-hospital mortality associated with traumatic brain injury in Canada: A nationwide, population-based study. J Trauma Acute Care Surg. 2015 Sep;79(3):449-54. doi: 10.1097/ta.0000000000000733. PMID 26535433
- [Background] Jiang R, Zhao S, Wang R, Feng H, Zhang J, Li X, Mao Y, Yuan X, Fei Z, Zhao Y, Yu X, Poon WS, Zhu X, Liu N, Kang D, Sun T, Jiao B, Liu X, Yu R, Zhang J, Gao G, Hao J, Su N, Yin G, Zhu X, Lu Y, Wei J, Hu J, Hu R, Li J, Wang D, Wei H, Tian Y, Lei P, Dong JF, Zhang J. Safety and Efficacy of Atorvastatin for Chronic Subdural Hematoma in Chinese Patients: A Randomized ClinicalTrial. JAMA Neurol. 2018 Nov 1;75(11):1338-1346. doi: 10.1001/jamaneurol.2018.2030. PMID 30073290
- [Background] Kudo H, Kuwamura K, Izawa I, Sawa H, Tamaki N. Chronic subdural hematoma in elderly people: present status on Awaji Island and epidemiological prospect. Neurol Med Chir (Tokyo). 1992 Apr;32(4):207-9. doi: 10.2176/nmc.32.207. PMID 1378564
- [Background] Balser D, Farooq S, Mehmood T, Reyes M, Samadani U. Actual and projected incidence rates for chronic subdural hematomas in United States Veterans Administration and civilian populations. J Neurosurg. 2015 Nov;123(5):1209-15. doi: 10.3171/2014.9.JNS141550. Epub 2015 Mar 20. PMID 25794342
- [Background] Brennan PM, Kolias AG, Joannides AJ, Shapey J, Marcus HJ, Gregson BA, Grover PJ, Hutchinson PJ, Coulter IC; British Neurosurgical Trainee Research Collaborative. The management and outcome for patients with chronic subdural hematoma: a prospective, multicenter, observational cohort study in the United Kingdom. J Neurosurg. 2017 Mar 17:1-8. doi: 10.3171/2016.8.JNS16134.test. Online ahead of print. PMID 28306417
- [Background] Rauhala M, Helen P, Huhtala H, Heikkila P, Iverson GL, Niskakangas T, Ohman J, Luoto TM. Chronic subdural hematoma-incidence, complications, and financial impact. Acta Neurochir (Wien). 2020 Sep;162(9):2033-2043. doi: 10.1007/s00701-020-04398-3. Epub 2020 Jun 10. PMID 32524244
- [Background] Balser D, Rodgers SD, Johnson B, Shi C, Tabak E, Samadani U. Evolving management of symptomatic chronic subdural hematoma: experience of a single institution and review of the literature. Neurol Res. 2013 Apr;35(3):233-42. doi: 10.1179/1743132813Y.0000000166. PMID 23485050
- [Background] Lee KS. Natural history of chronic subdural haematoma. Brain Inj. 2004 Apr;18(4):351-8. doi: 10.1080/02699050310001645801. PMID 14742149
- [Background] Sahyouni R, Goshtasbi K, Mahmoodi A, Tran DK, Chen JW. Chronic Subdural Hematoma: A Historical and Clinical Perspective. World Neurosurg. 2017 Dec;108:948-953. doi: 10.1016/j.wneu.2017.09.064. Epub 2017 Sep 19. PMID 28935548
- [Background] Cofano F, Pesce A, Vercelli G, Mammi M, Massara A, Minardi M, Palmieri M, D'Andrea G, Fronda C, Lanotte MM, Tartara F, Zenga F, Frati A, Garbossa D. Risk of Recurrence of Chronic Subdural Hematomas After Surgery: A Multicenter Observational Cohort Study. Front Neurol. 2020 Nov 24;11:560269. doi: 10.3389/fneur.2020.560269. eCollection 2020. PMID 33329304
- [Background] Hammer A, Tregubow A, Kerry G, Schrey M, Hammer C, Steiner HH. Predictors for Recurrence of Chronic Subdural Hematoma. Turk Neurosurg. 2017;27(5):756-762. doi: 10.5137/1019-5149.JTN.17347-16.1. PMID 27593834
- [Background] Miranda LB, Braxton E, Hobbs J, Quigley MR. Chronic subdural hematoma in the elderly: not a benign disease. J Neurosurg. 2011 Jan;114(1):72-6. doi: 10.3171/2010.8.JNS10298. Epub 2010 Sep 24. PMID 20868215
- [Background] Weigel R, Schmiedek P, Krauss JK. Outcome of contemporary surgery for chronic subdural haematoma: evidence based review. J Neurol Neurosurg Psychiatry. 2003 Jul;74(7):937-43. doi: 10.1136/jnnp.74.7.937. PMID 12810784
- [Background] Liu W, Bakker NA, Groen RJ. Chronic subdural hematoma: a systematic review and meta-analysis of surgical procedures. J Neurosurg. 2014 Sep;121(3):665-73. doi: 10.3171/2014.5.JNS132715. Epub 2014 Jul 4. PMID 24995782
- [Background] Peng Z, Ban K, LeBlanc A, Kozar RA. Intraluminal tranexamic acid inhibits intestinal sheddases and mitigates gut and lung injury and inflammation in a rodent model of hemorrhagic shock. J Trauma Acute Care Surg. 2016 Aug;81(2):358-65. doi: 10.1097/TA.0000000000001056. PMID 27027557
- [Background] Adhiyaman V, Chatterjee I. Increasing incidence of chronic subdural haematoma in the elderly. QJM. 2017 Nov 1;110(11):775. doi: 10.1093/qjmed/hcx143. No abstract available. PMID 29025124
- [Background] Miki K, Abe H, Morishita T, Hayashi S, Yagi K, Arima H, Inoue T. Double-crescent sign as a predictor of chronic subdural hematoma recurrence following burr-hole surgery. J Neurosurg. 2019 Jan 4;131(6):1905-1911. doi: 10.3171/2018.8.JNS18805. Print 2019 Dec 1. PMID 30611142
- [Background] Feghali J, Yang W, Huang J. Updates in Chronic Subdural Hematoma: Epidemiology, Etiology, Pathogenesis, Treatment, and Outcome. World Neurosurg. 2020 Sep;141:339-345. doi: 10.1016/j.wneu.2020.06.140. Epub 2020 Jun 25. PMID 32593768
- [Background] van der Vlegel M, Spronk I, Oude Groeniger J, Toet H, Panneman MJM, Polinder S, Haagsma JA. Health care utilization and health-related quality of life of injury patients: comparison of educational groups. BMC Health Serv Res. 2021 Sep 19;21(1):988. doi: 10.1186/s12913-021-06913-3. PMID 34538243
- [Background] Matei VP, Rosca AE, Pavel AN, Paun RM, Gmel G, Daeppen JB, Studer J. Risk factors and consequences of traumatic brain injury in a Swiss male population cohort. BMJ Open. 2022 Jul 21;12(7):e055986. doi: 10.1136/bmjopen-2021-055986. PMID 35863843
- [Background] Lee KS. Chronic Subdural Hematoma in the Aged, Trauma or Degeneration? J Korean Neurosurg Soc. 2016 Jan;59(1):1-5. doi: 10.3340/jkns.2016.59.1.1. Epub 2016 Jan 20. PMID 26885279
- [Background] Almenawer SA, Farrokhyar F, Hong C, Alhazzani W, Manoranjan B, Yarascavitch B, Arjmand P, Baronia B, Reddy K, Murty N, Singh S. Chronic subdural hematoma management: a systematic review and meta-analysis of 34,829 patients. Ann Surg. 2014 Mar;259(3):449-57. doi: 10.1097/SLA.0000000000000255. PMID 24096761
- [Background] Bajsarowicz P, Prakash I, Lamoureux J, Saluja RS, Feyz M, Maleki M, Marcoux J. Nonsurgical acute traumatic subdural hematoma: what is the risk? J Neurosurg. 2015 Nov;123(5):1176-83. doi: 10.3171/2014.10.JNS141728. Epub 2015 May 8. PMID 25955872
- [Background] Miah IP, Tank Y, Rosendaal FR, Peul WC, Dammers R, Lingsma HF, den Hertog HM, Jellema K, van der Gaag NA; Dutch Chronic Subdural Hematoma Research Group. Radiological prognostic factors of chronic subdural hematoma recurrence: a systematic review and meta-analysis. Neuroradiology. 2021 Jan;63(1):27-40. doi: 10.1007/s00234-020-02558-x. Epub 2020 Oct 22. PMID 33094383
- [Background] Jang KM, Choi HH, Mun HY, Nam TK, Park YS, Kwon JT. Critical Depressed Brain Volume Influences the Recurrence of Chronic Subdural Hematoma after Surgical Evacuation. Sci Rep. 2020 Jan 24;10(1):1145. doi: 10.1038/s41598-020-58250-w. PMID 31980723
- [Background] Hutchinson PJ, Edlmann E, Bulters D, Zolnourian A, Holton P, Suttner N, Agyemang K, Thomson S, Anderson IA, Al-Tamimi YZ, Henderson D, Whitfield PC, Gherle M, Brennan PM, Allison A, Thelin EP, Tarantino S, Pantaleo B, Caldwell K, Davis-Wilkie C, Mee H, Warburton EA, Barton G, Chari A, Marcus HJ, King AT, Belli A, Myint PK, Wilkinson I, Santarius T, Turner C, Bond S, Kolias AG; British Neurosurgical Trainee Research Collaborative; Dex-CSDH Trial Collaborators. Trial of Dexamethasone for Chronic Subdural Hematoma. N Engl J Med. 2020 Dec 31;383(27):2616-2627. doi: 10.1056/NEJMoa2020473. Epub 2020 Dec 16. PMID 33326713
- [Background] Prud'homme M, Mathieu F, Marcotte N, Cottin S. A Pilot Placebo Controlled Randomized Trial of Dexamethasone for Chronic Subdural Hematoma. Can J Neurol Sci. 2016 Mar;43(2):284-90. doi: 10.1017/cjn.2015.393. Epub 2016 Feb 8. PMID 26853325
- [Background] Moskala M, Goscinski I, Kaluza J, Polak J, Krupa M, Adamek D, Pitynski K, Miodonski AJ. Morphological aspects of the traumatic chronic subdural hematoma capsule: SEM studies. Microsc Microanal. 2007 Jun;13(3):211-9. doi: 10.1017/S1431927607070286. PMID 17490504
- [Background] Yamashima T, Yamamoto S, Friede RL. [A comparative study of the capsular vessels of acute subdural hematoma in the chronic healing stage and those of chronic subdural hematoma]. Neurol Med Chir (Tokyo). 1983 Jun;23(6):428-36. doi: 10.2176/nmc.23.428. No abstract available. Japanese. PMID 6195537
- [Background] Kutty RK, Leela SK, Sreemathyamma SB, Sivanandapanicker JL, Asher P, Peethambaran A, Prabhakar RB. The Outcome of Medical Management of Chronic Subdural Hematoma with Tranexamic Acid - A Prospective Observational Study. J Stroke Cerebrovasc Dis. 2020 Nov;29(11):105273. doi: 10.1016/j.jstrokecerebrovasdis.2020.105273. Epub 2020 Sep 4. PMID 33066896
- [Background] Mebberson K, Colditz M, Marshman LAG, Thomas PAW, Mitchell PS, Robertson K. Prospective randomized placebo-controlled double-blind clinical study of adjuvant dexamethasone with surgery for chronic subdural haematoma with post-operative subdural drainage: Interim analysis. J Clin Neurosci. 2020 Jan;71:153-157. doi: 10.1016/j.jocn.2019.08.095. Epub 2019 Sep 3. PMID 31492485
- [Background] Giuffre R. Physiopathogenesis of chronic subdural hematomas: a new look to an old problem. Riv Neurol. 1987 Sep-Oct;57(5):298-304. PMID 3328270
- [Background] Nomura S, Kashiwagi S, Ito H, Mimura Y, Nakamura K. Degradation of fibrinogen and fibrin by plasmin and nonplasmin proteases in the chronic subdural hematoma: evaluation by sodium dodecyl sulfate-polyacrylamide gel electrophoresis and immunoblot. Electrophoresis. 1993 Dec;14(12):1318-21. doi: 10.1002/elps.11501401202. PMID 8137796
- [Background] Miranda I, Collado-Sanchez A, Peregrin-Nevado I, Diaz-Martinez JV, Sanchez-Alepuz E, Miranda FJ. Use of topical tranexamic acid in primary total hip arthroplasty. Efficiency and safety. Our experience. Rev Esp Cir Ortop Traumatol (Engl Ed). 2020 Mar-Apr;64(2):114-119. doi: 10.1016/j.recot.2019.09.011. Epub 2019 Nov 10. English, Spanish. PMID 31722865
- [Background] Markwalder TM. Chronic subdural hematomas: a review. J Neurosurg. 1981 May;54(5):637-45. doi: 10.3171/jns.1981.54.5.0637. No abstract available. PMID 7014792
- [Background] O YM, Tsang SL, Leung GK. Fibrinolytic-Facilitated Chronic Subdural Hematoma Drainage-A Systematic Review. World Neurosurg. 2021 Jun;150:e408-e419. doi: 10.1016/j.wneu.2021.03.029. Epub 2021 Mar 17. PMID 33722722
- [Background] McCormack PL. Tranexamic acid: a review of its use in the treatment of hyperfibrinolysis. Drugs. 2012 Mar 26;72(5):585-617. doi: 10.2165/11209070-000000000-00000. PMID 22397329
- [Background] Jawa RS, Singer A, Mccormack JE, Huang EC, Rutigliano DN, Vosswinkel JA. Tranexamic Acid Use in United States Trauma Centers: A National Survey. Am Surg. 2016 May;82(5):439-47. PMID 27215726
- [Background] Cai J, Ribkoff J, Olson S, Raghunathan V, Al-Samkari H, DeLoughery TG, Shatzel JJ. The many roles of tranexamic acid: An overview of the clinical indications for TXA in medical and surgical patients. Eur J Haematol. 2020 Feb;104(2):79-87. doi: 10.1111/ejh.13348. Epub 2019 Dec 16. PMID 31729076
- [Background] Yokobori S, Yatabe T, Kondo Y, Kinoshita K; Japan Resuscitation Council (JRC) Neuroresuscitation Task Force and the Guidelines Editorial Committee. Efficacy and safety of tranexamic acid administration in traumatic brain injury patients: a systematic review and meta-analysis. J Intensive Care. 2020 Jul 3;8:46. doi: 10.1186/s40560-020-00460-5. eCollection 2020. PMID 32637122
- [Background] Klebanoff JS, Marfori CQ, Ingraham CF, Wu CZ, Moawad GN. Applications of Tranexamic acid in benign gynecology. Curr Opin Obstet Gynecol. 2019 Aug;31(4):235-239. doi: 10.1097/GCO.0000000000000547. PMID 31022078
- [Background] Della Corte L, Saccone G, Locci M, Carbone L, Raffone A, Giampaolino P, Ciardulli A, Berghella V, Zullo F. Tranexamic acid for treatment of primary postpartum hemorrhage after vaginal delivery: a systematic review and meta-analysis of randomized controlled trials. J Matern Fetal Neonatal Med. 2020 Mar;33(5):869-874. doi: 10.1080/14767058.2018.1500544. Epub 2018 Sep 10. PMID 30122082
- [Background] Alanwar A, Abbas AM, Hussain SH, Elhawwary G, Mansour DY, Faisal MM, Elshabrawy A, Eltaieb E. Oral micronised flavonoids versus tranexamic acid for treatment of heavy menstrual bleeding secondary to copper IUD use: a randomised double-blind clinical trial. Eur J Contracept Reprod Health Care. 2018 Oct;23(5):365-370. doi: 10.1080/13625187.2018.1515349. Epub 2018 Sep 24. PMID 30247074
- [Background] WOMAN Trial Collaborators. Effect of early tranexamic acid administration on mortality, hysterectomy, and other morbidities in women with post-partum haemorrhage (WOMAN): an international, randomised, double-blind, placebo-controlled trial. Lancet. 2017 May 27;389(10084):2105-2116. doi: 10.1016/S0140-6736(17)30638-4. Epub 2017 Apr 26. PMID 28456509
- [Background] Khadanga P, Kanchi M, Gaur P. Effectiveness of Tranexamic Acid in Reducing Postoperative Blood Loss in Patients Undergoing Off-Pump Coronary Artery Bypass Grafting. Cureus. 2020 Dec 5;12(12):e11924. doi: 10.7759/cureus.11924. PMID 33425507
- [Background] Meissner F, Plotze K, Matschke K, Waldow T. Postoperative administration of tranexamic acid as approach to reduce blood loss after open-heart surgery. Clin Hemorheol Microcirc. 2020;76(1):43-49. doi: 10.3233/CH-200836. PMID 32417764
- [Background] Monaco F, Nardelli P, Pasin L, Barucco G, Mattioli C, Di Tomasso N, Dalessandro G, Giardina G, Landoni G, Chiesa R, Zangrillo A. Tranexamic acid in open aortic aneurysm surgery: a randomised clinical trial. Br J Anaesth. 2020 Jan;124(1):35-43. doi: 10.1016/j.bja.2019.08.028. Epub 2019 Oct 10. PMID 31607387
- [Background] Sprigg N, Flaherty K, Appleton JP, Al-Shahi Salman R, Bereczki D, Beridze M, Christensen H, Ciccone A, Collins R, Czlonkowska A, Dineen RA, Duley L, Egea-Guerrero JJ, England TJ, Krishnan K, Laska AC, Law ZK, Ozturk S, Pocock SJ, Roberts I, Robinson TG, Roffe C, Seiffge D, Scutt P, Thanabalan J, Werring D, Whynes D, Bath PM; TICH-2 Investigators. Tranexamic acid for hyperacute primary IntraCerebral Haemorrhage (TICH-2): an international randomised, placebo-controlled, phase 3 superiority trial. Lancet. 2018 May 26;391(10135):2107-2115. doi: 10.1016/S0140-6736(18)31033-X. Epub 2018 May 16. PMID 29778325
- [Background] Roberts I, Shakur-Still H, Aeron-Thomas A, Beaumont D, Belli A, Brenner A, Cargill M, Chaudhri R, Douglas N, Frimley L, Gilliam C, Geer A, Jamal Z, Jooma R, Mansukhani R, Miners A, Pott J, Prowse D, Shokunbi T, Williams J. Tranexamic acid to reduce head injury death in people with traumatic brain injury: the CRASH-3 international RCT. Health Technol Assess. 2021 Apr;25(26):1-76. doi: 10.3310/hta25260. PMID 33928903
- [Background] July J, Pranata R. Tranexamic acid is associated with reduced mortality, hemorrhagic expansion, and vascular occlusive events in traumatic brain injury - meta-analysis of randomized controlled trials. BMC Neurol. 2020 Apr 6;20(1):119. doi: 10.1186/s12883-020-01694-4. PMID 32252661
- [Background] Kozek-Langenecker SA, Ahmed AB, Afshari A, Albaladejo P, Aldecoa C, Barauskas G, De Robertis E, Faraoni D, Filipescu DC, Fries D, Haas T, Jacob M, Lance MD, Pitarch JVL, Mallett S, Meier J, Molnar ZL, Rahe-Meyer N, Samama CM, Stensballe J, Van der Linden PJF, Wikkelso AJ, Wouters P, Wyffels P, Zacharowski K. Management of severe perioperative bleeding: guidelines from the European Society of Anaesthesiology: First update 2016. Eur J Anaesthesiol. 2017 Jun;34(6):332-395. doi: 10.1097/EJA.0000000000000630. PMID 28459785
- [Background] Spahn DR, Bouillon B, Cerny V, Duranteau J, Filipescu D, Hunt BJ, Komadina R, Maegele M, Nardi G, Riddez L, Samama CM, Vincent JL, Rossaint R. The European guideline on management of major bleeding and coagulopathy following trauma: fifth edition. Crit Care. 2019 Mar 27;23(1):98. doi: 10.1186/s13054-019-2347-3. PMID 30917843
- [Background] Pagano D, Milojevic M, Meesters MI, Benedetto U, Bolliger D, von Heymann C, Jeppsson A, Koster A, Osnabrugge RL, Ranucci M, Ravn HB, Vonk ABA, Wahba A, Boer C. 2017 EACTS/EACTA Guidelines on patient blood management for adult cardiac surgery. Eur J Cardiothorac Surg. 2018 Jan 1;53(1):79-111. doi: 10.1093/ejcts/ezx325. No abstract available. PMID 29029100
- [Background] Kageyama H, Toyooka T, Tsuzuki N, Oka K. Nonsurgical treatment of chronic subdural hematoma with tranexamic acid. J Neurosurg. 2013 Aug;119(2):332-7. doi: 10.3171/2013.3.JNS122162. Epub 2013 May 3. PMID 23641825
- [Background] Lodewijkx R, Immenga S, van den Berg R, Post R, Westerink LG, Nabuurs RJA, Can A, Vandertop WP, Verbaan D. Tranexamic acid for chronic subdural hematoma. Br J Neurosurg. 2021 Oct;35(5):564-569. doi: 10.1080/02688697.2021.1918328. Epub 2021 Aug 2. PMID 34334070
- [Background] Wan KR, Qiu L, Saffari SE, Khong WXL, Ong JCL, See AA, Ng WH, King NKK. An open label randomized trial to assess the efficacy of tranexamic acid in reducing post-operative recurrence of chronic subdural haemorrhage. J Clin Neurosci. 2020 Dec;82(Pt A):147-154. doi: 10.1016/j.jocn.2020.10.053. Epub 2020 Nov 8. PMID 33317724
- [Background] Iorio-Morin C, Blanchard J, Richer M, Mathieu D. Tranexamic Acid in Chronic Subdural Hematomas (TRACS): study protocol for a randomized controlled trial. Trials. 2016 May 5;17(1):235. doi: 10.1186/s13063-016-1358-5. PMID 27150916
- [Background] Poulsen FR, Munthe S, Soe M, Halle B. Perindopril and residual chronic subdural hematoma volumes six weeks after burr hole surgery: a randomized trial. Clin Neurol Neurosurg. 2014 Aug;123:4-8. doi: 10.1016/j.clineuro.2014.05.003. Epub 2014 May 14. PMID 25012003
- [Background] Katayama K, Matsuda N, Kakuta K, Naraoka M, Takemura A, Hasegawa S, Akasaka K, Shimamura N, Itoh K, Asano K, Konno H, Ohkuma H. The Effect of Goreisan on the Prevention of Chronic Subdural Hematoma Recurrence: Multi-Center Randomized Controlled Study. J Neurotrauma. 2018 Jul 1;35(13):1537-1542. doi: 10.1089/neu.2017.5407. PMID 29444611
- [Background] Fujisawa N, Oya S, Yoshida S, Tsuchiya T, Nakamura T, Indo M, Matsui T. A Prospective Randomized Study on the Preventive Effect of Japanese Herbal Kampo Medicine Goreisan for Recurrence of Chronic Subdural Hematoma. Neurol Med Chir (Tokyo). 2021 Jan 15;61(1):12-20. doi: 10.2176/nmc.oa.2020-0287. Epub 2020 Nov 19. PMID 33208583
- [Background] Wang X, Song J, He Q, You C. Pharmacological Treatment in the Management of Chronic Subdural Hematoma. Front Aging Neurosci. 2021 Jul 1;13:684501. doi: 10.3389/fnagi.2021.684501. eCollection 2021. PMID 34276343
- [Background] Wu M, Wajeeh H, McPhail MN, Seyam O, Flora J, Nguyen H. Usage of Tranexamic Acid for Treatment of Subdural Hematomas. Cureus. 2023 Apr 15;15(4):e37628. doi: 10.7759/cureus.37628. eCollection 2023 Apr. PMID 37200656
- [Background] Immenga S, Lodewijkx R, Roos YBWEM, Middeldorp S, Majoie CBLM, Willems HC, Vandertop WP, Verbaan D. Tranexamic acid to prevent operation in chronic subdural haematoma (TORCH): study protocol for a randomised placebo-controlled clinical trial. Trials. 2022 Jan 18;23(1):56. doi: 10.1186/s13063-021-05907-0. PMID 35042560
- [Background] Alahmadi H, Vachhrajani S, Cusimano MD. The natural history of brain contusion: an analysis of radiological and clinical progression. J Neurosurg. 2010 May;112(5):1139-45. doi: 10.3171/2009.5.JNS081369. PMID 19575576
- [Background] Weng K, Zhang X, Bi Q, Zhao C. The effectiveness and safety of tranexamic acid in bilateral total knee arthroplasty: A meta-analysis. Medicine (Baltimore). 2016 Sep;95(39):e4960. doi: 10.1097/MD.0000000000004960. PMID 27684841
- [Background] Houston BL, Uminski K, Mutter T, Rimmer E, Houston DS, Menard CE, Garland A, Ariano R, Tinmouth A, Abou-Setta AM, Rabbani R, Neilson C, Rochwerg B, Turgeon AF, Falk J, Breau RH, Fergusson DA, Zarychanski R. Efficacy and Safety of Tranexamic Acid in Major Non-Cardiac Surgeries at High Risk for Transfusion: A Systematic Review and Meta-Analysis. Transfus Med Rev. 2020 Jan;34(1):51-62. doi: 10.1016/j.tmrv.2019.10.001. Epub 2019 Oct 23. PMID 31982293
- [Background] CRASH-2 Collaborators, Intracranial Bleeding Study. Effect of tranexamic acid in traumatic brain injury: a nested randomised, placebo controlled trial (CRASH-2 Intracranial Bleeding Study). BMJ. 2011 Jul 1;343:d3795. doi: 10.1136/bmj.d3795. PMID 21724564
- [Background] Uno M, Toi H, Hirai S. Chronic Subdural Hematoma in Elderly Patients: Is This Disease Benign? Neurol Med Chir (Tokyo). 2017 Aug 15;57(8):402-409. doi: 10.2176/nmc.ra.2016-0337. Epub 2017 Jun 26. PMID 28652561
- See also: Product Monograph for Marcan-Tranexamic Acid Tablets — https://pdf.hres.ca/dpd_pm/00066431.PDF
- See also: Related Info — https://www.healthmeasures.net/index.php?option=com_content&view=category&layout=blog&id=113&Itemid=808
- See also: Product Monograph for Sandoz-Tranexamic Acid Injection BP — https://pdf.hres.ca/dpd_pm/00066203.PDF